CLINICAL TRIAL: NCT03913546
Title: Acute Effects of Spinal Manipulation on the Neuromuscular Performance of Amateur Cyclists: Pilot Study
Brief Title: Spinal Manipulation and Neuromuscular Performance on Amateur Cyclists
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: In the first tests the force meter gave an error and all the records were lost. Then came the COVID-19 pandemic. At this time we are unable to finish the study. We hope to be able to complete it by the middle of next year.
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Francisco Germain, Associate professor, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CEI/HU/2018/09
Record Dates: First submitted 2019-04-04; First posted 2019-04-12 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Manual Therapies
Keywords: neuromuscular properties; strength; power; performance
MeSH Terms: interventions — Manipulation, Chiropractic

STUDY DESIGN:
Intervention Model Description: Randomized, parallel, pre-post study design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will receive either a sham procedure or the actual intervention. The researchers in charge of outcome assessment and statistical analysis will be blinded to the allocation of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham spinal manipulation (Sham Comparator): Participants in the 'sham' group will receive a sham mechanical thrust (force set at level 0) instead of an actual one. In the force level 0, no excursion of the stylus occurs, but the instrument produces the same clicking sound as in the actual SMT condition. Therefore, the subject does not distinguish between intervention or placebo.
  Interventions: Other: Sham spinal manipulative therapy
- Actual spinal manipulation (Experimental): Participants in the actual actual spinal manipulative therapy (SMT) group will be assessed through the Activator basic method. SMT will be performed with the Activator IV Adjusting Instrument (Activator Methods International, Phoenix, AZ) varying the force level depending on the adjusted segment.
  Interventions: Procedure: Spinal manipulative therapy

INTERVENTIONS:
Procedure: Spinal manipulative therapy — Participants in the actual spinal manipulative therapy group will be assessed through the activator basic method protocol. SMT will be performed with an Activator IV (Activator Methods International, Phoenix, AZ) setting the force at level 3 for the low thoracic spine (T7-T12), and level 4 for the lumbar spine and pelvis.
  Other Names: Chiropractic manipulation; Spine thrust manipulation
  Arms: Actual spinal manipulation
Other: Sham spinal manipulative therapy — Participants in the sham SMT group will undergo a protocol identical to the actual one, with the exception that a sham mechanical thrust (force set at level 0) will be delivered to the targeted areas. In the force level 0 no excursion of the stylus occurs, but the instrument produces the same clicking sound as in the actual SMT condition
  Arms: Sham spinal manipulation

SUMMARY:
The present study aims to assess the effects of spinal manipulation therapy on neuromuscular performance.

DETAILED DESCRIPTION:
The present study will follow a parallel, pre-post design. The aim will be to determine the acute effects of spinal manipulation therapy (SMT) on different neuromuscular properties of recreational cyclists. Specifically, the investigators will measure the maximum force production capacity and muscle activation of the knee extensors concomitantly during a maximal voluntary contraction, as well as the maximum and mean power attained during a Wingate cycling test (i.e., 30 seconds 'all out'). Participants will undergo the tests on two different occasions separated by at least 48 hours and a maximum of 2 weeks. The same tests will be conducted in both testing sessions, but participants will be randomly assigned into two groups (sham or actual SMT) immediately before the second testing session.

ELIGIBILITY:
Inclusion Criteria:

* Will be recruited from three different local triathlon and cycling clubs.
* Will have to cycle at least 4 hours per week during the preceding 3 months, and to have a cycling experience greater than 2 years

Exclusion Criteria:

* Having suffered an injury in the month before the study that precluded regular exercise practice
* Having suffered any type of spine injury before the study
* Having previously received Spinal Manipulation Therapy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Maximal force | On the control session and on the intervention session (immediately after the sham or actual SMT procedure)
  Peak force registered during an isometric maximal voluntary contraction of the knee extensors.
Voluntary activation | On the control session and on the intervention session (immediately after the sham or actual SMT procedure)
  Electromyographic activity of the vastus lateralis muscle registered during an isometric maximal voluntary contraction of the knee extensors.
Peak power | On the control session and on the intervention session (immediately after the sham or actual SMT procedure)
  Peak power registered during a 30-second Wingate anaerobic cycling test
Mean power | On the control session and on the intervention session (immediately after the sham or actual SMT procedure)
  Mean power registered during a 30-second Wingate anaerobic cycling test

CONTACTS AND LOCATIONS:
Overall Officials: Pedro de la Villa, MD, PhD, Study Director — University of Alcalá
Locations (1):
- University of Alcalá, Alcalá de Henares, Spain

REFERENCES:
- [Background] Valenzuela PL, Pancorbo S, Lucia A, Germain F. Spinal Manipulative Therapy Effects in Autonomic Regulation and Exercise Performance in Recreational Healthy Athletes: A Randomized Controlled Trial. Spine (Phila Pa 1976). 2019 May 1;44(9):609-614. doi: 10.1097/BRS.0000000000002908. PMID 30325889

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT03913546/Prot_SAP_000.pdf